CLINICAL TRIAL: NCT06058819
Title: Validation of Biomarkers Performance to Reduce Antibiotics overUse in newBorns With Suspected Clinical Signs of InfectionS
Acronym: RUBIS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0633
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Late Onset Sepsis
Keywords: neonatal sepsis,; biomarker; diagnostic,; antibiotic use; preterm neonates; NICU
MeSH Terms: conditions — Neonatal Sepsis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Newborns suspected of Infections — This study will include NICU newborns of at least 7 days of life with suggestive signs of neonatal sepsis. The results will be extrapolated to this same population.

SUMMARY:
Late-onset neonatal sepsis (LOS), occurring in newborn of at least 7 days of life, is frequently observed in Neonatal Intensive Care Units (NICUs) and potentially severe (mortality, neurologic and respiratory impairments).

Despite its high prevalence, a reliable diagnostic remains difficult. Currently, nonspecific clinical signs that might be related to other neonatal conditions such as prematurity and birth defects, are used to determine the diagnosis of LOS. Laboratory results of biological markers, such as C-Reactive Protein (CRP) and Procalcitonin (PCT) are often delayed in comparison with LOS onset. Blood culture results are too late and lack sensitivity. This explains why excessive antibiotic use is observed in a large proportion of NICU hospitalized newborns. This results in an increased antibiotic resistance, microbiota modification, neonatal complications (pulmonary, ophthalmologic and neurologic) and mortality.

A previous study (EMERAUDE) aimed to identify new biomarkers to early exclude the diagnosis of LOS, in order to limit antibiotic overuse. This study including 230 neonates revealed high performances of IL6, IL10, NGAL and combinations of PCT/IL10 and PTX3/NGAL.

The main objective of the present study will be to validate the performances of these biomarkers in another cohort. The secondary objectives will be to explore transcriptomic biomarkers and salivary biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the NICU of one of the two recruiting centers at the time of inclusion
* Patients aged ≥ 7 days
* Patients weighted ≥ 500 g the day of blood sample
* patients with suggestive signs of LOS including at least one of the following:Fever > 38°C; tachycardia > 160bpm; capillary refill time > 3 seconds; grey and/or pale skin complexion; apnea/ bradycardia syndrome, bloating; vomiting; rectal bleeding; hypotonia; lethargy; seizures without other obvious cause; increased ventilatory support and/or increased FiO2; cutaneous rash; inflammation at the needle-puncture site of the central venous catheter; or any other condition for which the clinician suspected an infection
* patients with a standard of care blood sampling, including at least a blood culture;

Exclusion Criteria:

* Patient treated with antibiotics for a bacteriologically confirmed infection at the time of sampling or within 48 hours prior to sampling
* Patient who underwent surgery within the previous 7 days
* Patients vaccinated within the previous 7 days
* Patient who received treatment with systemic corticosteroid therapy in the 48 hours prior to sampling
* Patient with severe combined immunodeficiency
* Opposition from parent(s)/guardian(s)

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns aged ≥ 7 days hospitalized in one of the 2 neonatal intensive care units (Nantes or Lyon) for whom an infection is suspected.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of late onset sepsis | 72 hours maximum after inclusion
  The primary outcome measure will be determined by an independent adjudication committee that will classify the patients into the following categories : infection, non infected or undetermined. This committee will be blinded to the biomarkers of the study. It will be composed of two neonatologists and a pediatrician specialized in pediatric infectious diseases.
  The diagnostic performance of the biomarkers combination will be based on the adjudication committee classification (gold standard).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - neonatal Intensive care unit, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, France, Bron
  - Hôpital Couple-Enfant - CHU Grenoble Alpes, Grenoble
  - Neonatal intensive care unit, Hôpital femme-maternité, Nantes

IPD SHARING:
Plan to Share IPD: No